CLINICAL TRIAL: NCT03033277
Title: Human Umbilical Cord Mesenchymal Stem Cells (HUC-MSCs) Transplantation in Women With Primary Ovarian Insufficiency (POI)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Hongmei Wang, Professor, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Multi-cited POI Recovery
Record Dates: First submitted 2017-01-10; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Hormone replacement therapy, placebo transplantation.
  Interventions: Biological: Placebo transplantation
- Experimental group (Experimental): Hormone replacement therapy,HUC-MSCs transplantation.
  Interventions: Biological: HUC-MSCs transplantation

INTERVENTIONS:
Biological: Placebo transplantation — Intraovarian injection of placebo through vagina under the guidance of ultrasonic.
  Arms: Control group
Biological: HUC-MSCs transplantation — Intraovarian injection of HUC-MSCs through vagina under the guidance of ultrasonic.
  Arms: Experimental group

SUMMARY:
There is a high incidence of women suffering from Primary Ovarian Insufficiency (POI). One of the most common treatments for POI is hormone replacement therapy (HRT), but HRT doesn't work well, and it has been shown to increase the risk of blood clots in the veins, ovarian cancer, and breast cancer. The ability of MSCs to differentiate into oocyte-like cells has been previously documented. Herein the purpose of this work is to evaluate the therapeutic potential of cell therapy in women suffering from POI.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary ovarian insufficiency;
2. Women between 20 and 40 years;
3. Have fertility requirements, husband has sperm;
4. Willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Primary amenorrhea;
2. Abnormal karyotyping (e.g. turner syndrome, fragile X syndrome);
3. Thyroid dysfunction;
4. Severe endometriosis;
5. Contraindications for pregnancy;
6. Prior personal history of ovarian cancer;
7. Unwilling to comply with follow-up schedule or want to take other treatment during the follow-up period;
8. History of serious drug allergy or allergic constitution;
9. Autoimmune disease, history of severe familial genetic disease;
10. HIV+, hepatitis B, C;

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of mature follicle | Up to 4 months
  The number of mature follicles developing was recorded by transvaginal ultrasound scan

SECONDARY OUTCOMES:
Follicle-stimulating hormone (FSH) serum level | Up to 4 months
  Serum FSH level was evaluated once a month after surgery
Estradiol (E2) serum level | Up to 4 months
  Serum E2 level was evaluated once a month after surgery
Anti-Mullerian hormone (AMH) serum level | Up to 4 months
  Serum AMH level was evaluated once a month after surgery
Number of antral follicle development | Up to 4 months
  The number of antral follicles developing was recorded by transvaginal ultrasound scan
Ovarian volume | Up to 4 months
  The ovarian volume was recorded by transvaginal ultrasound scan
Pregnancy rate | Up to 12 months
  The incidence of pregnancy following transfer of embryos produced from oocytes recovered from follicles developing was assessed by Serum Human Chorionic Gonadotropin (HCG) detection.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Wang, Doctor, Principal Investigator — State Key Laboratory of Stem Cell and Reproductive Biology
Locations (1):
- Institute of Zoology, Chinese Academy of Sciences., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No